CLINICAL TRIAL: NCT05963412
Title: Developing an Online Individual Intervention Program to Make Sense of People's Experiences After a Breast Cancer Diagnosis and Examining Its Effectiveness
Brief Title: Online Individual Intervention Program to Make Sense of People's Experiences After a Breast Cancer Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Selva Ülbe, Assistant Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeaningInt-BreastCancer
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; meaning making; online intervention program; psychological health
MeSH Terms: conditions — Breast Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Individual Intervention Program (Experimental): The online intervention program (namely, Meaning-Centered Coping Program) consists of eight individual sessions, each lasting approximately 60 min. Sessions were conducted per week.
  Interventions: Other: Meaning Centered Coping Program
- No Intervention: Waitlist Control Group (No Intervention): A wait-list control group was used. Participants assigned to the wait-list control group did not receive the intervention immediately. After the final assessment was administered (eight weeks later since the initial assessment), they were able to participate in the same intervention program if they wanted.

INTERVENTIONS:
Other: Meaning Centered Coping Program — Meaning Centered Coping Program is a psychological intervention program developed for women diagnosed with breast cancer, based on the Meaning Making Model (Park, 2010; Park and Folkman, 1997) and Wong's (2010) principles of Meaning Therapy. Each weekly session had specific topics. These are:
  Session 1: Guiding patients to tell the story of their breast cancer and psycho-education; Session 2: Encouraging patients to talk about the effects of breast cancer on their lives and learning to accept their difficult emotions; Session 3: Focusing on cognition through the meaning attributed to breast cancer; Session 4: Learning to take alternative perspectives and defusing their negative thoughts; Session 5: Exploring personal strengths; Session 6: İdentifying important life values and moving toward value-based actions; Session 7: Finding meaning in breast cancer and life; Session 8: Focusing on Future plans and hopes
  Arms: Online Individual Intervention Program

SUMMARY:
The unexpected changes caused by the diagnosis and treatment of breast cancer can lead individuals to question their beliefs, life meanings, and goals, prompting a search for meaning. According to Park and Folkman's Meaning-Making Model, the process of meaning making functions as a coping mechanism. It helps individuals adapt challenging experiences into their lives, ultimately assisting in their psychological adjustment to stressful situations. Based on this theoretical model, principles from meaning therapy literature reviews, interviews with breast cancer patients, and expert consultation, an 8-week online individual psychological intervention was developed. It was aimed at facilitating the finding of new meanings in the experience of breast cancer and promoting psychological well-being. It includes psycho-educational, cognitive, existential, and behavioral components explicitly focusing on the meaning-making process. This intervention is called the Meaning Centered Coping Program (MCCP). The main purpose of this study was to test whether the MCCP was an effective intervention program for women diagnosed with breast cancer. For this purpose, the study sample consisted of women with stage I, II, and III breast cancer. Then, participants were randomly assigned to the MCCP group and the waitlist control group. A number of reliable and valid measurement tools were used to compare the MCCP group with the waitlist control group and to examine the effect of the program. Compared with the control group, significant improvements were expected in the level of meaning in life, post-traumatic growth, situational meanings, and psychological well-being in the MCCP group.

DETAILED DESCRIPTION:
In recent years, there has been a growing discussion about the necessity for mental health services not only to alleviate individuals' psychological distress but also to focus on enhancing the sense of meaning in life. Therefore, the MCCP aimed not only to reduce distressing psychological symptoms but also to facilitate the discovery of new positive meanings in breast cancer and individual's life, despite existing limitations. In this regard, the MCCP has been developed by drawing upon Meaning-Making Model, principles of meaning therapy, the literature on meaning, and existing meaning centered psychotherapy approaches. Additionally, considering limitations such as potential program changes, transportation difficulties, and inadequate physical conditions, online interventions offer a reliable alternative that provides numerous advantages for individuals diagnosed with breast cancer. Therefore, the intervention program was implemented online via video conference for women diagnosed with breast cancer in the current study. After the program was developed, a pilot study was conducted. According to the expert's feedback, the final version of MCCP was developed. The primary aim was to test the effectiveness of MCCP among women with breast cancer. The research hypotheses are 1) compared to control grup, MCCP group would show better improvement in meaning in life and PTG scores 2) compared to control grup, MCCP group would show better improvements in situational meaning (i.e. stress appraisal 3)Compared to control group, the MCCP group would report a significantly lower level of psychological distress.

Before the data collection process, ethical approval was obtained from the Institutional Ethics Committee of Dokuz Eylül University, affiliated with Dokuz Eylül University School of Medicine (Ethics Committee Decision No: 2021/12-39). The study has been announced using social media platforms (Facebook, Twitter, Instagram), oncology associations established to support oncology patients, and referrals from healthcare professionals to reach potential participants. The sample size was determined using the power analysis method. Then, 44 women diagnosed with breast cancer who volunteered to participate in the study were randomly assigned to either the intervention group or the waitlist control group.

The random assignment process was conducted using the website https://www.randomizer.org/. Participants in the MCCP group were assessed thrice: before the intervention, immediately after the intervention, and at the 2-month follow-up. The control group underwent the initial assessment before intervention began and the final assessment took place eight weeks later. After getting verbal and written consent from all participants, a number of measurement tools was applied. The Sociodemographic and Disease-Related Information Form, The Meaning in Life Questionnaire, Posttraumatic Growth Inventory-X, Stress Appraisal Measure, and Hospital Anxiety and Depression Scale were used. To test the hypotheses of the study, Pearson correlation analysis, 2 (Group) X 2 (Time) repeated measures ANOVA, and one-way repeated measures ANOVA were applied. SPSS 29.0 Package Program for Social Sciences was used for statistical analyses.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 65 years
* Being a woman
* Being a native Turkish speaker
* Diagnosed with stage I, II, or III breast cancer
* Diagnosed for at least 6 months and at most 3 years
* Being able to video-conference using a desktop computer, a laptop, or a tablet

Exclusion criteria:

* Having any psychiatric diagnosis or currently using psychiatric medication,
* Currently receiving psychological support,
* Having a history of cancer diagnosis
* Having a diagnosis of advanced stage (stage ıv) breast cancer
* Having a concurrent diagnosis of another cancer.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study included women diagnosed with breast cancer. In this regard, biological sex was considered.
Enrollment: 44 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Socio-demographic and Disease-Related Information Form | Baseline (before the intervention program begins)
  This form is a questionnaire designed to gather socio-demographic characteristics and information related to the diagnosis of breast cancer from the participants. Socio-demographic questions include the participant's age, educational level, occupation, income level, marital status, the number of children, and health insurance coverage. The questions related to breast cancer include the time since diagnosis, clinical stage of breast cancer, duration of treatment, completed treatment, type of surgical interventions, cancer history and menstrual status.
Change in the Meaning in Life Questionnaire | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up
  The Meaning in Life Scale was developed to measure individuals' level of meaning and purpose in life (Steger et al., 2006) The scale consists of a total of ten items and comprises two dimensions: the presence of meaning and the search for meaning. The scale is assessed using a 7 point scale scored from 1 to 7. The Turkish version of The Meaning in Life Questionnaire, adapted by Akin and Taş (2015), was used in this study. Psychometric features of the Turkish version of the scale indicated that it was a valid and reliable measurement tool.
Change in Post-traumatic Growth Inventory-X | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The Posttraumatic Growth Inventory (PTGI) is developed to assess positive changes experienced following traumatic life events. In this study, the Posttraumatic Growth Inventory-X (PTGI-X) was used (Tedeschi et al., 2017). The inventory consists of 25 items and is scored on a six-point scale scored from 0 to 5. Higher scores on the inventory indicated higher levels of posttraumatic growth. The Psychometric properties of the inventory are sufficient to measure the level of post-traumatic growth.

SECONDARY OUTCOMES:
Change in The Stress Appraisal Measure | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The scale developed by Peacock and Wong (1990) is designed to assess the cognitive evaluation of stress. It consists of 24 items. The items are evaluated using a likert scale scored from 1 to 5. The scale comprises five subscales that involve primary (threat and challenge) and secondary appraisals (uncontrollable-by-anyone, controllable-by-self, and controllable-by-others). The scale is recommended by Park and George (2013) for assessing situational meaning. The Turkish version of the scale was used for this purpose in the current study.
Change in Global Meaning Violation Scale | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The scale developed by Park and colleagues (2016) is designed to assess disruptions in global meaning following a traumatic or stressful life event. It consists of 13 items. Each item of the scale is evaluated using a five-point scale scored from 1 to 5. Psychometric results demonstrated that the Turkish version of the scale was valid and reliable (Acet et al., 2020).
Change in The Impact of Event Scale-Revised | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The scale was developed to assess traumatic stress symptoms (Weiss,2004). It consists of 22 items, which are evaluated using a Likert scale scored from 0 to 4. The scale comprises three subscales. These are intrusion, avoidance, and hyperarousal . The adaptation of the scale to Turkish was conducted by Çorapçıoğlu and colleagues (2006). Within the scope of the current study, intrusions and avoidance were used to assess automatic meaning-making efforts.
Change in Acceptance and Action Questionnaire-II | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The Acceptance and Action Questionnaire-II (AAQ-II) was developed to measure psychological inflexibility/flexibility (Bond et al., 2011). The scale consists of a total of seven items, each of which is rated on a seven-point scale scored from 1 to 7. Higher scores on the scale indicate higher levels of psychological inflexibility. The scale has been adapted into Turkish by Meunier and colleagues (2014).Turkish version of the scale demonstrated adequate psychometric properties.
Change in The Hospital Anxiety and Depression Scale | Baseline (before the intervention program), post-intervention at 8 week (after the intervention program) and at the 2-month follow-up.
  The scale was developed by Zigmond and Snaith (1983) to assess the levels of depression and anxiety in individuals diagnosed with various physical illnesses. The scale consists of a total of 14 items, with seven items evaluating anxiety and another seven items assessing depression levels. Participants are asked to rate each item on a four-point scale ranging from 0 to 3. The Turkish validity and reliability study of the Hospital Anxiety and Depression Scale (HADS) was conducted by Aydemir and colleagues (1997). The HADS is a valid and reliable measurement tool for assessing anxiety and depression levels in samples with a medical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Selva Ülbe, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Faculty of Letters, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No